CLINICAL TRIAL: NCT06935994
Title: Aspirin for Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease: A Randomized Controlled Trial
Brief Title: Aspirin for Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF24404A
Record Dates: First submitted 2025-04-06; First posted 2025-04-20 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: This phase 2, double-blind, randomized, placebo-controlled trial will recruit MASLD patients, who fulfill the inclusion and exclusion criteria of this study, at Taichung Veterans General Hospital. Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo for 240 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin arm (Active Comparator): Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo
  Interventions: Drug: Aspirin 81 mg Enteric Coated Tab - 1 tablet
- Placebo arm (Placebo Comparator): Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin 81 mg Enteric Coated Tab - 1 tablet — Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo
  Other Names: Un-impede E.F.C.
  Arms: Aspirin arm
Drug: Placebo — Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo
  Other Names: Placebo Tablet
  Arms: Placebo arm

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is a leading cause of chronic liver disease worldwide and a significant public health issue. MASLD may progress to liver cirrhosis and/or hepatocellular carcinoma. Although previous evidence suggests that aspirin has antisteatotic and antifibrotic effects on the liver, a randomized controlled trial assessing long-term efficacy and safety of aspirin in MASLD patients has yet to be conducted. This study aims to conduct a randomized controlled trial to evaluate the efficacy of aspirin in treating MASLD.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) has become one of the most common chronic liver diseases, with an estimated prevalence exceeding 30% globally. MASLD can result in liver cirrhosis, hepatocellular carcinoma (HCC), and death, and it has become the leading cause of HCC waiting for liver transplantation in the U.S. Unfortunately, although several new drugs put forth in clinical trials have been shown to offer certain benefits towards improving MASLD, an effective medicine remains lacking. With the limitations in efficacy and safety issues, even though some medications maybe hopeful in the treatments for MASLD, more medical choices remain highly expected. Emerging laboratory evidence suggests that antiplatelet therapy, e.g., aspirin, can reduce the risk of MASLD progression; however, a well-designed clinical trial should be mandatory before its clinical use. A recently published 6-month, phase 2 randomized controlled trial (RCT) demonstrated that daily aspirin might improve MASLD, but several limitations of this study should be further investigated. Therefore, we aim to conduct a RCT to evaluate the long-term effect of low-dose aspirin therapy on MASLD. This phase 2, double-blind, randomized, placebo-controlled trial will recruit MASLD patients, who fulfill the inclusion and exclusion criteria of this study. Participants will be randomly assigned in a 1:1 ratio to receive daily low-dose (81mg) aspirin or a placebo for 240 weeks. Participants will be follow-up at outpatient clinics every 12 weeks, and liver stiffness measurement (LSM) will be evaluated by using vibration-controlled transient elastography (VCTE). The surrogate primary endpoint is mean absolute change of VCTE-estimated liver stiffness at week 48. The clinical- outcome primary endpoint is MASLD-related outcomes (LSM progression >= 5 kPa, liver decompensation, HCC development, cardiovascular events, and death) at week 240. The secondary endpoints include mean absolute changes of hepatic fat fraction measured by 1H-MR spectroscopy and liver function parameters and the cumulative incidence of bleeding events. Additionally, the study will explore associations between stool microbiota/ MASLD-related single nucleotide polymorphisms, such as PNPLA3, TM6SF2, MBOAT7 genes, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Diagnosed with MASLD, which is defined by the Delphi consensus, with at least one out of five cardiometabolic criteria

Exclusion Criteria:

1. Increased alcohol intake (average ≥ 20 g/day for women and ≥ 30 g/day for men)
2. Glycated hemoglobin (HbA1c) level ≥ 9.0%
3. Other causes of chronic liver disease, such as HBV, HCV, autoimmune hepatitis, Wilson's disease, etc.
4. Liver decompensation (Child-Pugh class B or C)
5. Liver cirrhosis with significant portal hypertension (platelet count < 100,000/mm3, splenomegaly, and/or the presence of esophageal/gastric varices)
6. High-risk EGV, defined as F2, F3, or with red-color signs, diagnosed by endoscopy within 6 months before screening
7. Active peptic ulcer disease diagnosed by endoscopy within 6 months be- fore screening
8. FIB-4 index < 1.3 at screening
9. Indicated for any anti-platelet therapy, such as history of cardiovascular events
10. History of aspirin allergy
11. History of bleeding disorders, such as hemophilia
12. Pregnancy or breast feeding
13. Severe renal impairment, which is defined as eGFR < 30 mL/min/1.73 m²
14. Any malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean absolute change of VCTE-estimated LSM | Week 48
  The surrogate primary endpoint is mean absolute change of VCTE-estimated LSM (kPa).
Cumulative incidence of MASLD-related clinical outcomes | Week 240
  The clinical-outcome primary endpoint is the cumulative incidence (%) of any MASLD-related adverse outcomes, including LSM progression >= 5 kPa, liver decompensation, HCC development, cardiovascular events, and death.

SECONDARY OUTCOMES:
Mean percentage change of VCTE-estimated LSM | Week 48, Week 240
  Mean percentage change of LSM measured by VCTE (%)
Changes in hepatic fat fraction | Week 48, Week 240
  Mean change of hepatic fat fraction measured by MRS (%)
Mean absolute changes of serum AST/ ALT | Week 48, Week 240
  Mean absolute changes of serum AST, ALT (U/L)
Mean percentage changes of serum AST/ ALT | Week 48, Week 240
  Mean percentage changes of serum AST/ ALT (%)

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, MBA, PhD, Study Chair — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No